CLINICAL TRIAL: NCT03983824
Title: A Phase 1 Study of M3814 in Combination With MEC in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Testing the Addition of an Anti-cancer Drug, M3814, to the Usual Treatment (Mitoxantrone, Etoposide, and Cytarabine) for Relapsed or Refractory Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-03607; NCI-2019-03607 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHI-103; 10273 (Other: City of Hope Comprehensive Cancer Center LAO); 10273 (Other: CTEP); UM1CA186717 (NIH)
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Specimen Handling; Biopsy; Cytarabine; etoposide phosphate; Mitoxantrone; peposertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (peposertib, mitoxantrone, etoposide, cytarabine) (Experimental): Patients receive peposertib PO BID on days 2-21, mitoxantrone IV over 15 minutes, etoposide IV over 60 minutes and cytarabine IV over 60 minutes on days 1-5 in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo ECHO or MUGA during baseline, and blood collection and bone marrow biopsy throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Drug: Cytarabine; Procedure: Echocardiography Test; Drug: Etoposide Phosphate; Drug: Mitoxantrone Hydrochloride; Procedure: Multigated Acquisition Scan; Drug: Peposertib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Etoposide Phosphate — Given IV
  Other Names: Etopophos
Drug: Mitoxantrone Hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Dihydroxyanthracenedione Dihydrochloride; Mitoxantrone Dihydrochloride; Mitoxantroni Hydrochloridum; Mitozantrone Hydrochloride; Mitroxone; Neotalem; Novantrone; Onkotrone; Pralifan
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Peposertib — Given PO
  Other Names: 3-Pyridazinemethanol, alpha-(2-Chloro-4-fluoro-5-(7-(4-morpholinyl)-4-quinazolinyl)phenyl)-6-methoxy-, (alphaS)-; M 3814; M-3814; M3814; MSC 2490484A; MSC-2490484A; MSC2490484A; Nedisertib

SUMMARY:
This phase I trial studies the best dose and side effects of M3814 when given in combination with mitoxantrone, etoposide, and cytarabine in treating patients with acute myeloid leukemia that has come back (relapsed) or does not respond to treatment (refractory). M3814 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as mitoxantrone and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Etoposide is in a class of medications known as podophyllotoxin derivatives. It blocks a certain enzyme needed for cell division and DNA repair and may kill cancer cells. Giving M3814 in combination with mitoxantrone, etoposide, and cytarabine may lower the chance of the acute myeloid leukemia growing or spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety and tolerability and determine the recommended phase two dose (RP2D) of peposertib (M3814) in combination with mitoxantrone, etoposide, and cytarabine (MEC) in patients with relapsed or refractory (R/R) acute myeloid leukemia (AML).

SECONDARY OBJECTIVES:

I. To characterize the pharmacokinetic (PK) profile of MEC alone and of M3814 in combination with MEC.

II. To evaluate the preliminary efficacy of M3814 in combination with MEC in patients with R/R AML as measured by the response rate (complete remission [CR] plus CR with incomplete count recovery [CRi]), duration of CR/CRi (DOR), event-free survival (EFS) and overall survival (OS).

EXPLORATORY OBJECTIVES:

I. To evaluate correlative biomarkers of M3814 target engagement and response. II. To correlate cytogenetic and molecular abnormalities with response. III. To evaluate the rates of early mortality and allogeneic hematopoietic cell transplantation.

IV. To perform molecular profiling assays on malignant and normal tissues, including, but not limited to, whole exome sequencing (WES) and messenger ribonucleic acid (RNA) sequencing (RNAseq), in order to:

IVa. Identify potential predictive and prognostic biomarkers beyond any genomic alteration by which treatment may be assigned; IVb. Identify resistance mechanisms using genomic deoxyribonucleic acid (DNA)- and RNA-based assessment platforms.

V. To contribute genetic analysis data from de-identified biospecimens to Genomic Data Commons (GDC), a well annotated cancer molecular and clinical data repository, for current and future research; specimens will be annotated with key clinical data, including presentation, diagnosis, staging, summary treatment, and if possible, outcome.

OUTLINE: This is a dose-escalation study of peposertib followed by a dose-expansion study.

Patients receive peposertib orally (PO) twice daily (BID) on days 2-21, mitoxantrone intravenously (IV) over 15 minutes, etoposide IV over 60 minutes and cytarabine IV over 60 minutes on days 1-5 in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo echocardiogram (ECHO) or multigated acquisition scan (MUGA) during baseline, and blood collection and bone marrow biopsy throughout the study.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 1 year, then every 6 months thereafter up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* An established and confirmed diagnosis of AML by World Health Organization criteria, excluding acute promyelocytic leukemia (APL) (with promyelocytic leukemia -retinoic acid receptor alpha [PML-RARA])
* Patients with R/R AML, defined as:

  * Relapsed: >= 5% bone marrow blasts by morphology, reappearance of peripheral blood blasts, or development of extramedullary leukemia after achieving prior CR or CRi. First or second relapse is eligible. First relapse is restricted to participants with CR 1 duration of less than 9-12 months
  * Refractory: no CR or CRi after one or more cycles of induction. Induction cycles include regimens with the intent to achieve remission and can include high intensity and/or low intensity regimens
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of M3814 in combination with mitoxantrone, etoposide, and cytarabine in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (or Karnofsky >= 60%)
* Serum bilirubin =< 1.5 institutional upper limit of normal (ULN) (For patients with hemolysis, Gilbert's syndrome or liver infiltration with leukemia, serum bilirubin =< 3 x institutional ULN)
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN (For patients with liver infiltration with leukemia, AST[SGOT]/ALT[SGPT] =< 5 x institutional ULN)
* Glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula
* Patients must be medically eligible to receive MEC, including acceptable pre-study cardiac function (left ventricular ejection fraction of >= 45%) and lifetime anthracycline exposure (=< 360 mg/m^2 daunorubicin equivalents)
* Patients may have had prior allogeneic hematopoietic cell transplant at least 3 months prior to enrollment but should not have evidence of active graft versus host disease or require systemic immune suppression
* Patients must be willing to submit the blood sampling and bone marrow sampling for any mandatory PK and pharmacodynamics analyses and exploratory biomarkers
* Female patients with child bearing potential must have a negative serum pregnancy test within 72 hours prior to the first study drug administration and all patients must be willing to use effective methods of contraception during the treatment period and 3 months after study completion
* Human immunodeficiency virus (HIV)-infected patients will be eligible for this trial if they are on effective antiretroviral regimens utilizing non-CYP-interacting agents, they have an undetectable viral load, they have a CD4 count > 350 cells/mm^3, and they have no history of acquired immune deficiency syndrome (AIDS)-defining opportunistic infections. If there is evidence of chronic hepatitis B virus (HBV) infection, HBV viral load must be undetectable on suppressive therapy, if indicated. If there is history of hepatitis C virus (HCV) infection, the patient must have been treated and have undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible
* All non-hematologic adverse events (AEs) of prior chemotherapy, surgery, or radiotherapy, except alopecia, must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade =< 1 prior to starting therapy

Exclusion Criteria:

* Patients must not have had prior treatment with MEC
* Patients must not have documented active central nervous system (CNS) involvement by leukemia. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events (AEs)
* Patients must not have received any other investigational or commercial agents or therapies administered with the intention to treat their leukemia within 14 days or 5 elimination half-lives (whichever is shorter) of first receipt of study drug, with the exception of hydroxyurea and/or leukapheresis used to control white blood cell counts
* Patients who cannot discontinue concomitant medications or herbal supplements that are strong inhibitors or strong inducers of cytochrome P450 (CYP) isoenzymes CYP3A4/5, CYP2C9 and CYP2C19 during treatment with M3814. Concomitant use of CYP1A2, CYP2B6 and CYP3A4/5 substrates with a narrow therapeutic index are also excluded during treatment with M3814. Patients may confer with the study doctor to determine if alternative medications can be used. The following categories of medications and herbal supplements must be discontinued for at least the specified period of time prior to the first dose of M3814:

  * Strong inducers of CYP3A4/5, CYP2C9 and CYP2C19: >= 3 weeks or 5 elimination half-lives (whichever is shorter) prior to the first dose of M3814
  * Strong inhibitors of CYP3A4/5, CYP2C9 and CYP2C19: >= 1 week or 5 elimination half-lives (whichever is shorter) prior to the first dose of M3814
  * Substrates of CYP1A2, CYP2B6 and CYP3A4/5 with a narrow therapeutic index: >= 1 day prior to the first dose of M3814
* Concomitant use of histamine-2 (H2)-blockers or proton pump inhibitors should be avoided as these might affect absorption of M3814; administrations have to be discontinued at least 5 days or 5 elimination half-lives (whichever is shorter) prior to the first dose of M3814. Antacid drugs should not be taken 1 hour before and until 2 hours after M3814 administration
* Patients receiving sorivudine or any chemically related analogues (such as brivudine) are excluded
* Patients who require oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes (including coumadin and warfarin), or who received such agents within 5 days or 5 elimination half-lives (whichever is shorter) of the first dose of M3814. Low and high-molecular weight heparins are permitted provided the platelets are maintained at greater than 30,000/mm^3
* Patients with ongoing active infection or who have received a live attenuated vaccine within 30 days of dosing with M3814
* Patients must not have known significant cardiopulmonary disease defined as:

  * Unstable angina;
  * Congestive heart failure (New York Heart Association [NYHA] class III or IV);
  * Myocardial infarction (MI) within 6 months prior to first dose. Patients who had ischemic heart disease such as acute coronary syndrome (ACS), MI, and/or revascularization more than 6 months before screening and who are without cardiac symptoms or those with a prior non-ST elevation MI (NSTEM) due to demand-supply mismatch (NSTEM Type II) may enroll
* Patients should not have severe and/or uncontrolled medical conditions or other conditions that, in the opinion of the investigator, could affect their participation in the study
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Patients should not be pregnant or breastfeeding
* A marked baseline prolongation of QT/corrected QT (QTc) interval (e.g., repeated demonstration of a QTc interval > 480 milliseconds [ms] [CTCAE grade 2] using Fredericia's QT correction formula)
* A history of additional risk factors for TdP (e.g., heart failure, hypokalemia, family history of Long QT syndrome)
* The use of concomitant medications that prolong the QT/QTc interval
* Gastrointestinal disorders that may affect the M3814 absorption
* Patients will need to avoid any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days before the first administration of M3814 and throughout the duration of M3814 treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 5 years
  Coded according to the Common Terminology Criteria for Adverse Events version 5.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile of M3814 in combination with mitoxantrone, etoposide, and cytarabine (MEC) | Days 1 and 5
  Individual PK parameters will be estimated for maximum concentration, area under the concentration-time curve, half-life, apparent clearance, and apparent volume of distribution using non-compartmental methods. The PK variables will be tabulated and descriptive statistics (e.g., geometric means and coefficients of variation) calculated for each dose level. PK parameters will be reported descriptively for exploratory comparison with historical data.
Overall response rate | Up to 5 years
  Defined as the proportion of subjects with complete remission (CR) plus CR with incomplete count recovery (CRi) using European Leukemia Net response criteria. The percent of CR will be calculated and associated exact 95% confidence intervals will be constructed.
Duration of CR/CRi | From first documented CR/CRi response to relapse, assessed up to 5 years
  Summarized using Kaplan-Meier plots.
Event-free survival | From study entry to treatment failure (lack of response, i.e., no CR or CRi), relapse from CR or CRi, or death from any cause, assessed up to 5 years
  Summarized using Kaplan-Meier plots.
Overall survival | From study entry to death from any cause, assessed up to 2 years
  Summarized using Kaplan-Meier plots.

OTHER OUTCOMES:
Rate of early mortality | At 90 days
  Defined as the proportion of subjects with death from any cause at 90 days after starting study treatment.
Rate of allogeneic hematopoietic cell transplantation (HCT) | Up to 5 years
  Defined as the proportion of subjects proceeding to allogeneic HCT after starting study treatment.
Pharmacodynamic effects of M3814 in combination with MEC | Up to 5 years
  Studies with pharmacodynamic (biological endpoints, toxicity and efficacy) will be analyzed using nonparametric statistics.
Effect of cytogenetic and molecular abnormalities | Baseline
  Will assess the effect of cytogenetic and molecular abnormalities as potential predictive biomarkers of sensitivity to these regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Jonas, Principal Investigator — City of Hope Comprehensive Cancer Center LAO
Locations (15):
- United States (15):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mount Sinai Hospital, New York, New York
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm